CLINICAL TRIAL: NCT05858684
Title: Dual Target CAR-T Cell Treatment for Refractory Systemic Lupus Erythematosus (SLE) Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Gracell Biotechnologies (Shanghai) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Qiong Fu, Professor, RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC012F-615
Record Dates: First submitted 2023-05-05; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: CAR-T Cell Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GC012F injection (CD19-BCMA CAR-T cells) (Experimental): Dose escalation phase:
  DL-1：0.5±20%×10^5/kg, DL1：1±20%×10^5/kg, DL2：2±20%×10^5/kg DL3：3±20%×10^5/kg
  Interventions: Drug: GC012F injection

INTERVENTIONS:
Drug: GC012F injection — Each subject will receive GC012F injection (CD19-BCMA CAR-T cells) by intravenous infusion on Day 0.
  Other Names: CD19-BCMA CAR-T cells

SUMMARY:
This is an early exploratory phase, single arm, non-randomized, open label, treatment study trial to determine the maximum tolerated dose of GC012F injection (CD19-BCMA CAR-T cells) in patients with refractory systemic lupus erythematosus.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a kind of autoimmune diseases mediated by autoantibody-forming immune complexes, which involving multiple systems and organs.

Autoreactive B cells can self-activate and differentiate into plasma cells releasing large amounts of autoantibodies, while they can also present their own antigens to autoimmune T cells, thus activating T cells and promoting the release of inflammatory factors.

Traditional SLE treatment aims at long-term remission, while, CD19- BCMA CAR-T cells can theoretically completely deplete abnormal antibody-producing B cells, allowing immune rebuilding and restoring the patient's normal immune function, achieving drug-free survival, which fully reflects the application prospects of CAR-T therapy in SLE.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old;
2. Total score ≥ 10 on the EULAR/ACR 2019 SLE classification criteria;
3. SELENA-SLEDAI≥8;
4. Patients with CD19+ B-cell;
5. Hemoglobin≥85 g/L;
6. WBC≥2.5×10^9/L
7. NEUT≥1×10^9/L;
8. BPC≥50×10^9/L;
9. AST/ALT below 2 times the upper limit of normal; Creatinine clearance ≥30 mL/min; blood bilirubin ≤2.0 mg/dl; echocardiography indicates that the ejection fraction is ≥50%;
10. Adequate venous access for apheresis, and no other contraindications for leukapheresis;
11. Women of childbearing age should have a negative serum or urine pregnancy test at screening and baseline. Subjects agree to take effective contraceptive measures during the trial until at least 1 year after CAR-T cells infusion.
12. Agree to attend follow-up visits as required;
13. Voluntary participation and informed consent signed by the patient or his/her legal/authorized representative;

Exclusion Criteria:

1. Renal disease: severe lupus nephritis (serum creatinine > 2.5 mg/dL or 221 μmol/L) within 8 weeks prior to leukapheresis, or subjects who need hemodialysis;
2. CNS disease: including epilepsy, psychosis, organic encephalopathy syndrome, cerebrovascular accident [CVA], encephalitis or CNS vasculitis, psychiatric patients with depression or suicidal thoughts;
3. Patients with serious lesions and history of present illness of vital organs such as heart, liver, kidney and blood and endocrine system;
4. Patients with immunodeficiency, uncontrolled active infections and active or recurrent peptic ulcers;
5. Received immunosuppressive therapy within 1 week prior to leukapheresis;
6. Patients with HIV infection; Active infection of hepatitis B virus or hepatitis C virus; Patients with syphilis infection;
7. The presence or suspicion of an active fungal, bacterial, viral or other infection that cannot be controlled during screening;
8. Received live vaccine treatment within 4 weeks prior to screening;
9. Severe allergies or hypersensitivity;
10. Contraindication to cyclophosphamide in combination with fludarabine;
11. Subjects who have undergone major surgery within 2 weeks prior to signing the informed consent form, or who are scheduled to have surgery (other than local anesthetic surgery) during the trial or within 2 weeks of the infusion;
12. cannula or drainage tubes other than central venous catheters;
13. Pregnant or lactating women, or subjects who plan to have children within 1 year of treatment;
14. Subjects with prior CD19 or BCMA-targeted therapy
15. Participated in any clinical study within 3 months prior to enrollment
16. Subjects with malignant tumour, except for Non-melanoma Skin Cancer with PFS>5yr; Cervical Cancer in situ; Bladder Cancer; Breast Cancer;
17. Any situations that the investigator believes the patients are not suitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-05-11 (Estimated); Primary Completion 2023-11-10 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with DLT | Within 28 days after GC012F injection infusion
  DLT definition is dose-limiting toxicity
The proportion of subjects with adverse events | Within 12 weeks after GC012F injection infusion
  All adverse events were evaluated according to NCI-CTCAE v5.0 criteria

SECONDARY OUTCOMES:
Proportion of subjects achieving SRI-4 | 4, 8, 12 and 24 weeks after GC012F injection infusion
  SELEAN-SLEDAI，BILAG，PGA
Number of CAR-T cells and CAR gene copies in subjects'blood and bone marrow (if applicable) | After GC012F injection infusion [day 4, 7, 10, 14 and week 4, 8, 12, 24]
  Test method: flow cytometry and qPCR

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rheumatology, Ren Ji Hospital South Campus, School of Medicine, Shanghai JiaoTong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No